CLINICAL TRIAL: NCT03615677
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Active-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of LXI-15028 Comparing With Esomeprazole in the Treatment of Erosive Esophagitis in Chinese Patients for up to 8 Weeks
Brief Title: Efficacy and Safety of LXI-15028 Comparing With Esomeprazole in the Treatment of Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC821602
Record Dates: First submitted 2018-07-09; First posted 2018-08-06 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Erosive Esophagitis (EE)
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LXI-15028 50mg group (n=130) (Experimental)
  Interventions: Drug: LXI-15028 50mg
- Esomeprazole 40mg group (n=130) (Active Comparator)
  Interventions: Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: LXI-15028 50mg — The investigational products are administrated orally, once in the morning every day, and each dose includes 2 tablets of investigational products (LXI-15028 50mg active agent + Esomeprazole 40mg matching placebo . If the investigational product is not taken in the morning, subjects can take it before 6:00 p.m. on the same day. The duration of treatment is 4 or 8 weeks.
  Arms: LXI-15028 50mg group (n=130)
Drug: Esomeprazole 40mg — The investigational products are administrated orally, once in the morning every day, and each dose includes 2 tablets of investigational products ( LXI-15028 50mg matching placebo + Esomeprazole 40mg active agent ). If the investigational product is not taken in the morning, subjects can take it before 6:00 p.m. on the same day. The duration of treatment is 4 or 8 weeks.
  Arms: Esomeprazole 40mg group (n=130)

SUMMARY:
This is a multi-center, randomized, double-blind, parallel-group, active controlled Phase III clinical study to evaluate the efficacy and safety of LXI-15028 50 mg comparing with esomeprazole 40 mg after the treatment of erosive esophagitis in Chinese patients for up to 8 weeks.

Screening-eligible subjects will be randomized into LXI-15028 50mg treatment group or esomeprazole 40mg treatment group at Visit 2 (Day 0) stratified by LA grade (A or B/C/D) at baseline according to the ratio of 1:1 and receive study treatment continuously for 4 or 8 weeks. They will start to take the investigational products from the following morning (Day 1) of Visit 2, and start to complete the subject's diary from the day of study treatment initiation. After 4 weeks of study treatment (treatment period 1), subjects will return to the study site and complete Visit 3. For the subjects who achieve endoscopic healing at Visit 3, the study treatment will be terminated. The subjects who fail to achieve endoscopic healing at Visit 3 will receive newly dispensed investigational product after completing the fasting examinations at Visit 3, and continue another 4 weeks of study treatment (treatment period 2) and complete Visit 4. All the subjects will be followed up by phone (Visit 5) at Day 28±3 after the last dose of investigational products.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subject who volunteers to sign the written informed consent form approved by the independent ethics committee and agrees to participate in this study prior to the initiation of any study procedures.

  2) Subject who is able to understand and comply with the protocol requirements and agrees to participate in all the study visits.

  3) Male or female subjects with age ≥ 18 years. 4) Having experienced heartburn and regurgitation within 7 days prior to screening, with the frequency and severity in symptom assessment meeting at least one of the following items:
* Mild heartburn for at least 2 days, with regurgitation;
* Mild regurgitation for at least 2 days, with heartburn;
* Moderate or more severe heartburn for at least 1 day, with regurgitation;
* Moderate or more severe regurgitation for at least 1 day, with heartburn. (Note: To be determined by using the RDQ [item a, b, e, f] completed by subject.) 5) Subject who is diagnosed as Los Angeles (LA) grade A to D erosive esophagitis through upper gastrointestinal endoscopy within 14 days prior to the initiation of study treatment. (Note: The target of enrollment is to ensure the number of subjects with LA grade A does not exceed 60% of the total number of subject enrolled)

Exclusion Criteria:

* 1) Subject who had participated in this study previously, or had participated in other P-CAB drug clinical studies.

  2) Participation in other clinical study within 3 months prior to screening, except for the two following circumstances:
* The study which the subject is participating or participated in is a non-interventional study (e.g. observational study or questionnaire survey) and is judged by investigators to have no interference with the efficacy and safety evaluation in the present study;
* Subject had signed the informed consent form and participated in another study (NC821603) sponsored by this sponsor in the same study site, but had been withdrawn from that study prior to the start of any treatment.

  3) Subjects who participate in the plan or conduction of this study (e.g., staff of the sponsor or study site).

  4) Subject who is known to be allergic to the active ingredient or excipient of the investigational product (including esomeprazole).

  5) Subject who is unable to undertake an upper gastrointestinal endoscopy. 6) Subject who is unable to complete the subject's diary by oneself. 7) Subject who has history of manic-depression, anxiety disorder, panic disorder, somatoform disorder, personality disorder or other mental disorder.

  8) Subject who has symptoms such as odynophagia, serious dysphagia, bleeding, decreased body weight, anemia or hematochezia that represent "warning" to presume gastrointestinal malignant disease, unless the possibility of the malignant disease is excluded through an endoscopy.

  9) Subject who is diagnosed as achalasia of the cardia, secondary esophageal motility disorder, irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), Zollinger-Ellison syndrome or eosinophilic esophagitis.

  10) Subject with history of digestive tract surgery, except for simple fenestration, appendectomy, cholecystectomy or endoscopic resection of benign tumor. 11) Subject who plans to be hospitalized for receiving selective surgery during the study.

  12) Subject with non-reflux-related esophageal stenosis, hiatus hernia, gastroesophageal varices, active peptic ulcer, gastric bleeding or malignant tumor that is found in upper gastrointestinal endoscopy.

  13) Subject with uncontrolled and unstable hepatic, renal, cardiovascular, respiratory, endocrine or central nervous system disease as judged by investigators.

  14) Subject with history of chronic alcohol consumption (more than 14 cups per week, each cup corresponds to 360 mL beer or 150 mL wine or 45 mL liquor) or drug abuse within 5 years prior to screening.

  15) Use of any PPI, P-CAB or other drugs related to the treatment of GERD (including H2-receptor antagonist, prostaglandin or mucosal protective agent), or any other antiemetic, emetic drugs within two weeks prior to the initiation of study treatment.

  16) Subject who needs non-steroidal anti-inflammatory drugs (NSAIDs) during the study, unless the subject had started to use low dose aspirin (≤ 100 mg/day) prior to screening.

  17) Use of potent-to-moderate cytochrome metabolism enzyme CYP3A4 inhibitor or inducer within 4 weeks prior to study treatment, including but not limited to the following drugs:
* CYP3A4 inhibitors: Ketoconazole, Indinavir, Saquinovir, Atazanavir, Amprenavir, Fosamprenavir, Nefazodone, Itraconazole, Telithromycin, Fluconazole, Troleandomycin, Cimetidine, Aprepitant, Fluvoxamine, Amiodarone, Ritonavir, Erythromycin, Clarithromycin, and Diltiazem;
* CYP3A4 inducers: Barbiturate, Phenytoin, Rifampin, St John's wort, Carbamazepine, Dexamethasone, Rifabutin, and Phenobarbital etc.; 18) Subject currently using antipsychotic drug, antidepressant agent or anti-anxiety agent.

  19) Any of the following laboratory abnormalities at screening:
* AST ≥ 2 x upper limit of normal (ULN);
* ALT ≥ 2 x ULN;
* ALP ≥ 2 x ULN;
* γ-GT ≥ 2 x ULN;
* Total bilirubin ≥ 2 x ULN;
* BUN (or urea) ≥ 1.5 x ULN;
* Creatinine ≥ 1.5 x ULN 20) Subject with clinically significant abnormality in ECG at screening, including serious arrhythmia, multifocal premature ventricular contraction (PVC), second degree or above atrioventricular block, prolonged QT interval (QTc ≥ 450 ms for male, QTc ≥ 470 ms for female).

  21) Current infection of human immune deficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) confirmed by tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Cumulative endoscopic healing rate | 4 or 8 weeks after receiving oral doses
  Percentage of patients with healing erosion based on the upper Gastrointestinal (GI) endoscopy following 8 weeks of study treatment

SECONDARY OUTCOMES:
Endoscopic healing rate at Week 4 | 4 week after receiving oral doses
  Percentage of patients with healing erosion based on the upper Gastrointestinal (GI) endoscopy following 4 weeks of study treatment
Change of Reflux Disease Questionnaire (RDQ) score for main symptoms | 4 or 8 weeks after receiving oral doses
  Total score for main symptoms (heartburn and regurgitation) (Total score is the sum of the score of heartburn and regurgitation, the range is 0-20, the higher score indicates the worse sympotom)
Change of Reflux Disease Questionnaire (RDQ) score for subcategory | 4 or 8 weeks after receiving oral doses
  Score for each Reflux Disease Questionnaire (RDQ) subcategory (heartburn, regurgitation and dyspepsia) (The range is 0-10 for every subcategory score)
Symptom assessment based on subject diary | 4 or 8 weeks after receiving oral doses
  Percentage of days without main symptoms (heartburn and regurgitation) during 1 week (7 days), 4 weeks and 8 weeks from the initiation of study treatment
Change of Gastro Esophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) score | 4 or 8 weeks after receiving oral doses
  Change of Gastro Esophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) score of each post-treatment visit from baseline at each post-treatment visit from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Doctor, Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhu H, Xue Q, Song Y, Zhang Z, Li X, Lyu S, Zhan Q, Liu F, Lu L, Zhong L, Chen W, Shao D, Ding Y, Liu D, Yang X, Huang Z, Li Z, Du Y. Efficacy and safety of tegoprazan (LXI-15028) vs. esomeprazole in patients with erosive esophagitis: A multicenter, randomized, double-blind, non-inferiority phase Ⅲ trial. Chin Med J (Engl). 2024 Oct 30;138(19):2464-71. doi: 10.1097/CM9.0000000000003276. Online ahead of print. PMID 39474720